CLINICAL TRIAL: NCT04866251
Title: Prevalence of Gag Reflex in Healthy Persons and Across Different Patient Groups and Its Relevance in Dysphagia Screening
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Giessen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Gag Reflex - 1
Record Dates: First submitted 2020-11-18; First posted 2021-04-29 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Neurological Diseases or Conditions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Healthy young subject (Active Comparator): Testing of gag reflex in different oral areas (tongue, velum, pharyngeal wall) and evaluation of present reactions. The Mallampati score is assessed in order to evaluate the feasibility of gag reflex test in case of higher Mallampati scores.
  Interventions: Diagnostic Test: Gag reflex test; assessment of Mallampati Score
- Healthy older subjects (Active Comparator): Testing of gag reflex in different oral areas (tongue, velum, pharyngeal wall) and evaluation of present reactions. The Mallampati score is assessed in order to evaluate the feasibility of gag reflex test in case of higher Mallampati scores.
  Interventions: Diagnostic Test: Gag reflex test; assessment of Mallampati Score
- Acute stroke patients (Active Comparator): Testing of gag reflex in different oral areas (tongue, velum, pharyngeal wall) and evaluation of present reactions. The Mallampati score is assessed in order to evaluate the feasibility of gag reflex test in case of higher Mallampati scores.
  Interventions: Diagnostic Test: Gag reflex test; assessment of Mallampati Score
- Patients with Parkinson´s Disease (Active Comparator): Testing of gag reflex in different oral areas (tongue, velum, pharyngeal wall) and evaluation of present reactions. The Mallampati score is assessed in order to evaluate the feasibility of gag reflex test in case of higher Mallampati scores.
  Interventions: Diagnostic Test: Gag reflex test; assessment of Mallampati Score
- Patients with Multiple Sclerosis (Active Comparator): Testing of gag reflex in different oral areas (tongue, velum, pharyngeal wall) and evaluation of present reactions. The Mallampati score is assessed in order to evaluate the feasibility of gag reflex test in case of higher Mallampati scores.
  Interventions: Diagnostic Test: Gag reflex test; assessment of Mallampati Score
- Patients with Myasthenia gravis (Active Comparator): Testing of gag reflex in different oral areas (tongue, velum, pharyngeal wall) and evaluation of present reactions. The Mallampati score is assessed in order to evaluate the feasibility of gag reflex test in case of higher Mallampati scores.
  Interventions: Diagnostic Test: Gag reflex test; assessment of Mallampati Score
- Geriatric patients (Active Comparator): Testing of gag reflex in different oral areas (tongue, velum, pharyngeal wall) and evaluation of present reactions. The Mallampati score is assessed in order to evaluate the feasibility of gag reflex test in case of higher Mallampati scores.
  Interventions: Diagnostic Test: Gag reflex test; assessment of Mallampati Score

INTERVENTIONS:
Diagnostic Test: Gag reflex test; assessment of Mallampati Score — Testing of gag reflex Assessment of Mallampati Score

SUMMARY:
The aim of this study is to assess the prevalence of gag reflex in healthy young and healthy older subjects as well as in acute stroke patients, in patients with Parkinsons´s Disease, Myasthenia gravis, Multiple Sclerosis and in geriatric patients.

DETAILED DESCRIPTION:
In the clinical swallowing examination in acute stroke setting it is assumed that the absence of gag reflex is a predictor of aspiration risk. According to Daniels et al. (1997) aspiration can be predicted with 96% sensitivity in case of absent or abnormal gag reflex. In clinical experience of investigators testing of gag reflex highly depends on patients´compliance and individual anatomical features such as Mallampati score. Furthermore, even if gag reflex is absent, swallowing does not have to be impaired.

The presence of gag reflex in healthy cohorts and dysphagic patients has been examined in a few studies. Davies et al. (1995) have shown that in 37% of healthy volunteers gag reflex was absent. Ramsey et al. (2005) have shown that approx. 89% of the patients without gag reflex had dysphagia and 31% without dysphagia had a gag reflex. In both studies it was not stated to what extent the gag reflex could be examined in case of a high Mallampati score.

The present study aims at assessing the prevalence of gag reflex in healthy and neurological cohorts. The study protocol foresees testing of gag reflex in different oral areas (tongue, velum, pharyngeal wall) and evaluating present reactions. The Mallampati score is assessed in order to evaluate the feasibility of gag reflex test in case of higher Mallampati scores.

All patients are tested once by one examiner.

ELIGIBILITY:
Inclusion Criteria:

* informed consent

Exclusion Criteria:

1. Healthy participants:

   Neurological diseases Pre-diagnosed dysphagia Percutaneous endoscopic gastrostomy (PEG) tube Head and neck tumours Chemo- and/or radiotherapy in the head and neck area Reflux disease Chronic obstructive pulmonary disease (COPD) Previous surgeries on the cervical spine or thyroid gland Vocal cord paresis
2. Geriatric patients Neurologic diseases
3. Stroke patients Head and neck tumours Chemo- and/or radiotherapy in the head and neck area Reflux disease COPD Previous surgeries on the cervical spine or thyroid gland Vocal cord paresis
4. Neurologic patients without stroke Head and neck tumours (except of intracranial tumors= Chemo- and/or radiotherapy in the head and neck area Reflux disease COPD Previous surgeries on the cervical spine or thyroid gland Vocal cord paresis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2016-08-10 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of gag reflex | Baseline
  Prevalence of gag reflex

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Braun, MD, Principal Investigator — University Hospital Giessen and Marburg, Campus Giessen
Locations (1):
- University Hospital Giessen and Marburg, Giessen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No